CLINICAL TRIAL: NCT07214675
Title: The Edison System for Treatment of Benign Prostatic Hyperplasia (BPH) Using Histotripsy
Acronym: WOLVERINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP5895
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: This is a prospective multi-center, single-arm, feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HistoSonics Edison System (Experimental)
  Interventions: Device: HistoSonics Edison System

INTERVENTIONS:
Device: HistoSonics Edison System — The HistoSonics Edison System is intended for the non-invasive mechanical destruction of prostate tissue for the treatment of BPH using histotripsy, a non-thermal, mechanical process of focused ultrasound.
  Other Names: Histotripsy

SUMMARY:
The purpose of this trial is to evaluate the safety of histotripsy using the HistoSonics Edison System for treatment of BPH.

DETAILED DESCRIPTION:
This is a prospective multi-center, single-arm, feasibility trial designed to evaluate the safety of the HistoSonics Histotripsy System for treatment of BPH. Following histotripsy, subjects will undergo imaging ≤ 72 hours post-index procedure. Additionally, subjects will be followed at 30-day, 90-day and 180-day timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 50 years of age.
2. Subject has signed the Ethics Committee (EC) approved trial Informed Consent Form (ICF) prior to any trial related tests/procedures and is willing to comply with trial procedures and required follow-up assessments.
3. Subject is diagnosed with BPH.
4. Subject has a Body Mass Index (BMI) < 27.
5. Subject has an I-PSS ≥ 15.
6. Subject has a prostate volume > 30 mL and ≤ 150 mL.
7. Subject has a Qmax ≤ 15 mL/s with a voided volume of ≥ 125 mL during a uroflow test.
8. Subject accepts the potential loss of ejaculatory function.
9. Subject can tolerate general anesthesia. Index-Procedure Imaging Inclusion (Assessed day of procedure)
10. Subject has an adequate acoustic window to visualize the prostate using the HistoSonics Edison System.
11. Target treatment volume is ≥ 1 cm from the rectum as visualized on ultrasound, CT or MR imaging.

Exclusion Criteria:

1. Subject has a life expectancy of less than one (1) year.
2. Subject has a known sensitivity to contrast media and cannot be adequately pre-medicated.
3. Subject has a post-void residual ≥ 150 mL confirmed via ultrasound.
4. Subject has an estimated glomerular filtration rate (eGFR) ≤ 50 mL/min, ≤ 14 days prior to the planned index procedure date.
5. Subject has uncorrectable coagulopathy.
6. Subject has an International Normalized Ratio (INR) value ˃ 2.0, ≤14 days prior to the planned index procedure date.
7. Subject has had a prostatectomy.
8. Subject has acute prostatitis.
9. Subject has a diagnosis of or has received treatment for chronic prostatitis or chronic pelvic pain syndrome.
10. Subject has had a urinary tract infection (UTI) ≤ 3 months prior to the planned index procedure date.
11. Subject has bladder stones.
12. Subject is catheter dependent or has a history of intermittent self-catheterization.
13. Presence of prostatic calcifications in the planned treatment volume (PTV).
14. Presence of permanent radioactive implants in the rectal wall.
15. Subject has has a major abdominal or rectal surgery that inhibits visualization of the prostate.
16. Subject has undergone prior locoregional therapy (e.g., Rezum, laser, Urolift, TURP emboli, or radiation).
17. Subject has planned locoregional therapy 6 months post index procedure (e.g., Rezum, laser, Urolift, TURP emboli, or radiation).
18. Subjects who have active cancers (not in remission for the last two years) other than non-melanomatous skin cancers.
19. Subject is being actively treated in another pharmaceutical or device trial that has not completed its primary endpoint prior to the index procedure or may interfere with the primary outcome measure of this trial.
20. In the investigator's opinion, histotripsy is not a treatment option for the subject.
21. Subject has a concurrent condition that could jeopardize the safety of the subject or compliance with the protocol.
22. Subject's prostate is not treatable by the System's working ranges (refer to User Guide).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of Index-Procedure Related Adverse Events Classified by Clavien-Dindo Classification and Common Terminology Criteria for Adverse Events (CTCAE) | 30 days post histotripsy procedure
  Index procedure-related complications ≤30 days post index procedure, graded using Clavien-Dindo Classification and Common Terminology Criteria for Adverse Events (CTCAE). [Clinical Events Committee Adjudicated]

IPD SHARING:
Plan to Share IPD: No